CLINICAL TRIAL: NCT05446870
Title: A Randomized, Phase 2 Study of Pembrolizumab And Chemotherapy With or Without MK-4830 as Neoadjuvant Treatment for High-Grade Serous Ovarian Cancer
Brief Title: Pembrolizumab With Chemotherapy and MK-4830 for Treating Participants With Ovarian Cancer (MK-4830-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4830-002; MK-4830-002 (Other: MSD); 2023-505005-16-00 (Registry Identifier: EU CT); U1111-1290-6634 (Registry Identifier: UTN); 2021-005458-27 (EudraCT Number)
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: High-grade Serous Ovarian Carcinoma; Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Paclitaxel; Carboplatin; Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Standard of Care (SOC) + MK-4830 (Experimental): Before surgery participants will receive pembrolizumab 200 mg, paclitaxel 175 mg/m^2 (or docetaxel 75 mg/m^2), carboplatin Area Under the Curve (AUC) 5 to 6, and MK-4830 800 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks [Q3W]) for 3 cycles. After surgery participants will receive pembrolizumab 200 mg, paclitaxel 175 mg/m^2 (or docetaxel 75 mg/m^2), carboplatin AUC 5 to 6, and MK-4830 800 mg (with avastin [or biosimilar] at the investigator's discretion and per insitutional guidelines) by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Biological: Avastin; Biological: MK-4830; Drug: Docetaxel
- Pembrolizumab + SOC (Active Comparator): Before surgery participants will receive pembrolizumab 200 mg, paclitaxel 175 mg/m^2 (or docetaxel 75 mg/m^2), and carboplatin AUC 5 to 6 by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles. After surgery participants will receive pembrolizumab 200 mg, paclitaxel 175 mg/m^2 (or docetaxel 75 mg/m^2), and carboplatin AUC 5 to 6 (with avastin [or biosimilar] at the investigator's discretion and per insitutional guidelines) by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Biological: Avastin; Drug: Docetaxel

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg by IV infusion on Day 1 of each 21-day cycle
  Other Names: MK-3475; KEYTRUDA®
Drug: Paclitaxel — 175 mg/m^2 by IV infusion on Day 1 of each 21-day cycle
  Other Names: TAXOL®
Drug: Carboplatin — AUC 5 to 6 by IV infusion on Day 1 of each 21-day cycle
  Other Names: PARAPLATIN®
Biological: Avastin — According to local practice and at the choice of the investigator.
  Other Names: Bevacizumab; Zirabev; MVASI; AYBINTIO; Versavo; Onbevezy; OYAVAS; ALYMSYS; Avegra
Biological: MK-4830 — 800 mg by IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab + Standard of Care (SOC) + MK-4830
Drug: Docetaxel — 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle

SUMMARY:
The primary objective is to evaluate in participants with high-grade serous ovarian cancer (HGSOC), whether the reduction from baseline in circulating tumor deoxyribonucleic acid (ctDNA) at Cycle 3 (ΔctDNA) is larger in participants receiving MK-4830 + pembrolizumab in combination with standard of care (SOC) therapy than in those receiving pembrolizumab + SOC therapy.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically-confirmed International Federation of Gynecology and Obstetrics (FIGO) Stage III or Stage IV HGSOC, primary peritoneal cancer, or fallopian tube cancer.
* Is a candidate for carboplatin and paclitaxel chemotherapy, to be administered in the neoadjuvant and adjuvant setting.
* Is a candidate for interval debulking surgery.
* Is able to provide archival tissue or newly obtained core, incisional, or excisional biopsy of a tumor lesion.
* Has adequate organ functions.

Exclusion Criteria:

* Has a non-HGSOC histology.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Has received prior treatment for any stage of ovarian cancer (OC), including radiation or systemic anticancer therapy.
* Planned or has been administered intraperitoneal chemotherapy as first-line therapy.
* Has received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-programmed cell death 1 ligand 1 (PD-L1), anti-programmed cell death 1 ligand 2 (PD-L2), anti-immunoglobulin-like transcript 4 (ILT4), or anti-human leukocyte antigen (HLA)-G agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity to pembrolizumab, carboplatin, paclitaxel (or docetaxel, if applicable), Avastin or biosimilar (if using) and/or any of their excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B or known active hepatitis C virus infection.
* Has received colony-stimulating factors within 4 weeks prior to receiving study intervention on Day 1 of Cycle 1.
* Has had surgery <6 months prior to Screening to treat borderline ovarian tumors, early-stage OC, or early-stage fallopian tube cancer.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has current, clinically relevant bowel obstruction.
* Has a history of hemorrhage, hemoptysis, or active gastrointestinal (GI) bleeding within 6 months prior to randomization.
* Has uncontrolled hypertension.
* Has had an allogenic tissue/solid organ transplant.
* Has either had major surgery within 3 weeks of randomization or has not recovered from any effects of any major surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with advanced high-grade serous ovarian cancer (HGSOC), fallopian tube cancer, or primary peritoneal cancer.
Enrollment: 160 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (45):
- United States (12):
  - University of Colorado Anschutz Medical Campus-Cancer Clinical Trials Office ( Site 0108), Aurora, Colorado
  - Mayo Clinic in Florida ( Site 0101), Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc. ( Site 0110), Miami, Florida
  - Northwestern Memorial Hospital ( Site 0104), Chicago, Illinois
  - Washington University ( Site 0113), St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey ( Site 0114), New Brunswick, New Jersey
  - Roswell Park Cancer Institute ( Site 0106), Buffalo, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0116), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone ( Site 0107), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0102), New York, New York
  - Sanford Cancer Center-Gynecologic Oncology ( Site 0115), Sioux Falls, South Dakota
  - Fred Hutchinson Cancer Center ( Site 0100), Seattle, Washington
- Belgium (3):
  - Antwerp University Hospital-Oncology ( Site 1301), Edegem, Antwerpen
  - AZ Maria Middelares-IKG ( Site 1302), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 1300), Leuven, Vlaams-Brabant
- Canada (2):
  - Centre Hospitalier de l'Université de Montréal ( Site 0300), Montreal, Quebec
  - McGill University Health Centre ( Site 0301), Montreal, Quebec
- Chile (4):
  - FALP ( Site 0905), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Centro del Cáncer ( Site 0900), Santiago, Region M. de Santiago
  - James Lind Centro de Investigación del Cáncer ( Site 0903), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0904), Viña del Mar, Región de Valparaíso
- Israel (3):
  - Rambam Health Care Campus-Gyneco-oncology unit ( Site 0602), Haifa
  - Shaare Zedek Medical Center ( Site 0601), Jerusalem
  - Sheba Medical Center-ONCOLOGY ( Site 0600), Ramat Gan
- Italy (4):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Oncologia Sperimentale Uro-Genitale ( Site 0, Napoli, Campania
  - Fondazione Policlinico Universitario Agostino Gemelli-Ginecologia Oncologica ( Site 0502), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Chirurgia Ginecologica ( Site 050, Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Ginecologia Oncologica ( Site 0501), Milan
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Poznaniu-Oddzial Ginekologii Onkologicznej ( Site 0709), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 0701), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Ginekologii Onkologicznej ( Sit, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Ginekologii, Ginekologii Onkologicznej i Endokrynologii Gi, Gdansk, Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej ( Site 0708), Kielce, Świętokrzyskie Voivodeship
- Singapore (2):
  - National Cancer Centre Singapore ( Site 1501), Singapore, Central Singapore
  - National University Hospital ( Site 1502), Singapore, South West
- South Korea (2):
  - Seoul National University Hospital ( Site 0801), Seoul
  - Severance Hospital, Yonsei University Health System-Gynecologic cancer center ( Site 0800), Seoul
- Spain (3):
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Medical Oncology ( Site 1103), Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 1104), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 1101), Barcelona
- Taiwan (5):
  - Changhua Christian Hospital-Obstetrics and Gynecology ( Site 1203), Changhua County, Changhua
  - Taichung Veterans General Hospital-GYNECOLOGY ( Site 1202), Taichung
  - National Cheng Kung University Hospital ( Site 1201), Tainan
  - National Taiwan University Hospital-Internal Medicine ( Site 1200), Taipei
  - Mackay Memorial Hospital ( Site 1204), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26295&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Standard of Care (SOC) + MK-4830: Before surgery participants received pembrolizumab, paclitaxel (or docetaxel), carboplatin, and MK-4830 by intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks [Q3W]) for 3 cycles. After surgery participants received pembrolizumab, paclitaxel (or docetaxel), and carboplatin (with avastin [or biosimilar] at the investigator's discretion and per institutional guidelines) by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles.
- Pembrolizumab + SOC: Before surgery participants received pembrolizumab, paclitaxel (or docetaxel), and carboplatin by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles. After surgery participants received pembrolizumab, paclitaxel (or docetaxel), and carboplatin (with avastin [or biosimilar] at the investigator's discretion and per institutional guidelines) by IV infusion on Day 1 of each 21-day cycle (Q3W) for 3 cycles.
Period: Overall Study
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Started | 80 | 80
Treated | 79 | 80
Completed | 19 | 18
Not Completed | 61 | 62
Not completed — Death | 6 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 52 | 53
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (9.5) | 61.5 (10.2) | 60.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 63 | 68 | 131
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 24 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 66 | 54 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Detectable Baseline Circulating Tumor Deoxyribonucleic Acid (ctDNA) [Mean (Standard Deviation); unit: MTM/mL] — Participants' blood samples were assessed at baseline for ctDNA mean mutant/tumor molecules per mL (MTM/mL). Population: Only participants with detectable ctDNA at baseline were included.
  MTM/mL
    number analyzed (Participants) | 64 | 68 | 132
    (all) | 214.4 (421.9) | 233.9 (393.2) | 224.5 (405.9)

OUTCOME MEASURES:

1. Secondary Outcome: Participants With Surgery and Pathological Complete Response (pCR): Change From Baseline in ctDNA
Description: Blood samples were collected to determine levels of ctDNA. pCR was defined as all surgical specimens collected during the interval debulking surgery microscopically negative for residual tumor. Per protocol, change from baseline in ctDNA in participants with surgery and pCR was reported.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least one dose of study intervention, had surgery, and had pCR and ctDNA data available for assessment.
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 39 | 53
Fold Change | 0.05 (0.13) | 0.04 (0.10)

2. Secondary Outcome: Association of Change From Baseline in ctDNA With pCR
Description: Blood samples were collected to determine levels of ctDNA. pCR was defined as all surgical specimens collected during the interval debulking surgery microscopically negative for residual tumor. pCR rate was defined as percentage of participants with pCR. Per protocol, the association of change from baseline in ctDNA with pCR in participants with surgery and pCR was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 39 | 53
Percentage of Participants | 12.8 [4.3 to 27.4] | 11.3 [4.3 to 23.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) + MK-4830 vs Pembrolizumab + SOC; Test type: Other; Posterior probability (%) = 100.00; Posterior probability (based on 20000 sets of model parameters) ctDNA fold change (square root scale) coefficient less than zero in the multivariable logistic regression model of pCR, adjusted for baseline ctDNA and treatment assignment

3. Secondary Outcome: Participants With Surgery and Chemotherapy Response Score (CRS): Change From Baseline in ctDNA
Description: Blood samples were collected to determine levels of ctDNA. CRS is a 3-tiered scoring system (CRS1-3) based on the pathological analysis of surgically removed omental masses. CRS was defined as CRS1 (minimal or no tumor response, mainly viable tumor), CRS2 (appreciable tumor response amidst viable tumor that is readily identifiable and regularly distributed), and CRS3 (complete or near-complete response, characterized by the lack of residual tumor cells in the omentum or presence of tumor foci up to 2 mm maximum size); higher values indicate greater response. Per protocol, change from baseline in ctDNA in participants with surgery and CRS was reported.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least one dose of study intervention, had surgery, and had CRS and ctDNA data available for assessment.
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 35 | 52
Fold Change | 0.09 (0.28) | 0.04 (0.10)

4. Secondary Outcome: Association of Change From Baseline in ctDNA With CRS3
Description: Blood samples were collected to determine levels of ctDNA. CRS is a 3-tiered scoring system (CRS1-3) based on the pathological analysis of surgically removed omental masses. CRS was defined as CRS1 (minimal or no tumor response, mainly viable tumor), CRS2 (appreciable tumor response amidst viable tumor that is readily identifiable and regularly distributed), and CRS3 (complete or near-complete response, characterized by the lack of residual tumor cells in the omentum or presence of tumor foci up to 2 mm maximum size); higher values indicate greater response. CRS3 rate was defined as percentage of participants with CRS3. Per protocol, the association of change from baseline in ctDNA with CRS3 in participants with surgery and CRS was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 35 | 52
Percentage of Participants | 45.7 [28.8 to 63.4] | 23.1 [12.5 to 36.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) + MK-4830 vs Pembrolizumab + SOC; Test type: Other; Posterior probability (%) = 90.99; Posterior probability (based on 20000 sets of model parameters) ctDNA fold change (square root scale) coefficient less than zero in the multivariable logistic regression model of CRS (CRS3 coded as 1 and CRS1 or 2 coded as 0), adjusted for baseline ctDNA and treatment assignment

5. Secondary Outcome: pCR Rate
Description: pCR rate was defined as the percentage of participants with all surgical specimens collected during the interval debulking surgery that were microscopically negative for residual tumor. The pCR rate as assessed by local pathologist was reported.
Time Frame: Up to approximately 12 weeks
Population: All randomized participants who received at least one dose of study intervention, received surgery, and had pCR data available for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 58 | 65
Percentage of Participants | 10.3 [3.9 to 21.2] | 9.2 [3.5 to 19.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) + MK-4830 vs Pembrolizumab + SOC; Test type: Other — Difference in percentage (calculated as % Pembrolizumab + SOC + MK-4830 arm - % Pembrolizumab + SOC arm) and 95% confidence interval (CI) were based on Miettinen & Nurminen method; Difference in Percentage = 1.1, 95% CI 2-sided [-10.0 to 12.9]

6. Secondary Outcome: CRS3 Rate
Description: CRS is a 3-tiered scoring system (CRS1-3) based on the pathological analysis of surgically removed omental masses. CRS was defined as CRS1 (minimal or no tumor response, mainly viable tumor), CRS2 (appreciable tumor response amidst viable tumor that is readily identifiable and regularly distributed), and CRS3 (complete or near-complete response, characterized by the lack of residual tumor cells in the omentum or presence of tumor foci up to 2 mm maximum size); higher values indicate greater response. CRS3 rate was defined as percentage of participants with CRS3. Per protocol, CRS3 rate as assessed by local pathologist was reported.
Time Frame: Up to approximately 12 weeks
Population: All randomized participants who received at least one dose of study intervention, received surgery, and had CRS data available for assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 55 | 61
Percentage of Participants | 43.6 [30.3 to 57.7] | 23.0 [13.2 to 35.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) + MK-4830 vs Pembrolizumab + SOC; Test type: Other — Difference in percentage (calculated as % Pembrolizumab + SOC + MK-4830 arm - % Pembrolizumab + SOC arm) and 95% CI were based on Miettinen & Nurminen method; Difference in Percentage = 20.7, 95% CI 2-sided [3.5 to 37.0]

7. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). The number of participants who experienced one or more AEs was reported.
Time Frame: Up to approximately 26 months
Population: All randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 79 | 80
Participants | 77 | 80

8. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated). The number of participants who discontinued study intervention due to an AE was reported.
Time Frame: Up to approximately 28 weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 79 | 80
Participants | 13 | 15

9. Primary Outcome: Change From Baseline in Circulating Tumor Deoxyribonucleic Acid (ctDNA)
Description: Blood samples were collected to determine levels of ctDNA. The fold change in the mean mutant/tumor molecules per mL (MTM/mL) at Cycle 3 from baseline is presented.
Time Frame: Baseline and Week 7
Population: All randomized participants who received at least one dose of study intervention, had detectable ctDNA at baseline, and had assessed ctDNA at Cycle 3.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
Number analyzed (Participants) | 51 | 63
Fold change | 0.08 (0.24) | 0.04 (0.10)
Statistical Analysis 1: Comparison: Pembrolizumab + Standard of Care (SOC) + MK-4830 vs Pembrolizumab + SOC; Test type: Other; Posterior probability (%) = 38.75; Posterior probability (based on 20000 sets of model parameters) coefficient for treatment assignment (MK-4830 containing vs. not) less than zero in Bayesian parametrization of the constrained longitudinal data analysis (cLDA) model, modeling ctDNA value at Cycle 3 and ctDNA value at baseline as bivariate normal

ADVERSE EVENTS:
Time Frame: Up to approximately 26 months
Description: All-Cause Mortality included all randomized participants. Serious and Other adverse events (AEs) included all randomized participants who received at least one dose of study intervention. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study intervention. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study intervention were excluded.
Arm/Group | Pembrolizumab + Standard of Care (SOC) + MK-4830 | Pembrolizumab + SOC
All-Cause Mortality (participants affected / at risk) | 6/80 | 5/80
Serious Adverse Events (participants affected / at risk) | 28/79 | 33/80
Other Adverse Events (participants affected / at risk) | 75/79 | 79/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Standard of Care (SOC) + MK-4830 (N=79) | Pembrolizumab + SOC (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (4)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superior mesenteric artery syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Serositis (General disorders) | 1 (1) | 0 (0)
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (2) | 1 (1)
Peritoneal abscess (Infections and infestations) | 1 (3) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Standard of Care (SOC) + MK-4830 (N=79) | Pembrolizumab + SOC (N=80)
Anaemia (Blood and lymphatic system disorders) | 44 (57) | 53 (92)
Leukopenia (Blood and lymphatic system disorders) | 14 (34) | 12 (16)
Neutropenia (Blood and lymphatic system disorders) | 21 (47) | 19 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (16) | 11 (14)
Hyperthyroidism (Endocrine disorders) | 4 (4) | 6 (6)
Hypothyroidism (Endocrine disorders) | 9 (9) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 19 (21) | 19 (29)
Constipation (Gastrointestinal disorders) | 29 (38) | 24 (30)
Diarrhoea (Gastrointestinal disorders) | 15 (19) | 19 (24)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 30 (36) | 35 (47)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 8 (8)
Vomiting (Gastrointestinal disorders) | 11 (16) | 18 (23)
Asthenia (General disorders) | 16 (29) | 20 (21)
Fatigue (General disorders) | 20 (23) | 16 (17)
Oedema peripheral (General disorders) | 4 (4) | 5 (5)
Pyrexia (General disorders) | 11 (13) | 12 (17)
Drug hypersensitivity (Immune system disorders) | 3 (4) | 5 (7)
COVID-19 (Infections and infestations) | 4 (4) | 9 (9)
Urinary tract infection (Infections and infestations) | 8 (9) | 13 (16)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 13 (14) | 21 (21)
Alanine aminotransferase increased (Investigations) | 9 (10) | 13 (16)
Aspartate aminotransferase increased (Investigations) | 8 (9) | 16 (20)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 9 (10)
Lymphocyte count decreased (Investigations) | 4 (7) | 9 (11)
Neutrophil count decreased (Investigations) | 11 (20) | 21 (41)
Platelet count decreased (Investigations) | 8 (11) | 21 (30)
Weight decreased (Investigations) | 6 (6) | 12 (13)
White blood cell count decreased (Investigations) | 6 (14) | 13 (20)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 13 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 16 (27)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 11 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (17) | 17 (26)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (9) | 11 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 11 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (20) | 11 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (17) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5) | 5 (6)
Dysgeusia (Nervous system disorders) | 5 (8) | 6 (10)
Headache (Nervous system disorders) | 7 (7) | 8 (10)
Neuropathy peripheral (Nervous system disorders) | 20 (20) | 28 (37)
Neurotoxicity (Nervous system disorders) | 4 (4) | 4 (6)
Paraesthesia (Nervous system disorders) | 7 (9) | 3 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 9 (9)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 10 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 35 (36) | 39 (40)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (14) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 15 (20) | 23 (30)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (10)
Hot flush (Vascular disorders) | 0 (0) | 6 (6)
Hypertension (Vascular disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT05446870/Prot_SAP_000.pdf